CLINICAL TRIAL: NCT07061899
Title: The Prevalence of Chlamydia Trachomatis and Neisseria Gonorrhoeae in Patients Suspected of Hemorrhagic Proctosigmoiditis
Acronym: SOSProctitis
Status: Active, not recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Regional Hospital Randers (Unknown); Central Jutland Regional Hospital (Other); Gødstrup Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SOS Proctitis
Record Dates: First submitted 2025-06-04; First posted 2025-07-11 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Proctitis, Ulcerative; Sexually Transmitted Disease (STD); Ulcerative Proctosigmoiditis
Keywords: Proctitis, Ulcerative; Ulcerative Proctosigmoiditis; Chlamydia trachomatis; Neisseria gonorrhoeae; Sexually Transmitted Diseases
MeSH Terms: conditions — Proctitis; Ulcer; Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Newly diagnosed haemorrhagic proctitis: First-ever episode, endoscopically confirmed within the specified enrolment window.
  Interventions: Diagnostic Test: Anal swap for Chlamydia and Gonorrhoea
- Recurrent haemorrhagic proctitis: One or more prior confirmed episodes and current relapse confirmed endoscopically.
  Interventions: Diagnostic Test: Anal swap for Chlamydia and Gonorrhoea

INTERVENTIONS:
Diagnostic Test: Anal swap for Chlamydia and Gonorrhoea — If inflammation is observed on endoscopy up to 35 cm from the anal opening, a swab will be taken during the procedure to test for Chlamydia and Gonorrhoea using standard PCR techniques. If the swab is not taken during the endoscopy, it will be collected during a follow-up outpatient visit. The tests will be analysed immediately at the Department of Microbiology, Aarhus University Hospital.
  If positve, the patient will be offered treatment at the department of Venerological diseases.

SUMMARY:
Background Chlamydia trachomatis and Neisseria gonorrhoeae can cause infectious proctitis, which macroscopically cannot be distinguished from haemorrhagic proctosigmoiditis (HP) caused by inflammatory bowel disease. In Denmark, general practitioners are advised to consider whether patients presenting with proctitis symptoms might have a sexually transmitted infection (STI). However, there is no requirement for STI testing before referring the patient to a specialised department.

At specialised departments, it is not standard practice to systematically inquire about sexual risk behaviour or to test for Chlamydia and Gonorrhoea. As a result, there is no data on how many patients diagnosed with HP due to chronic inflammatory bowel disease are also positive for an STI, either as the sole cause or as a contributing factor to their inflammation. Chlamydia and Gonorrhoea are the most common causes of symptomatic, sexually transmitted proctitis and are increasingly prevalent in Denmark.

Materials and methods Since diagnosing haemorrhagic proctosigmoiditis requires an endoscopy (sigmoidoscopy or colonoscopy), all newly diagnosed patients will undergo such an examination. Moreover, an endoscopy is often performed in individuals with refractory proctosigmoiditis. If inflammation is observed up to 35 cm from the anal opening, an additional swab will be taken during the procedure to test for Chlamydia and Gonorrhoea using standard PCR techniques. If the swab is not taken during the endoscopy, it will be collected during a follow-up outpatient visit. The tests will be analysed immediately at the Department of Microbiology, Aarhus University Hospital.

Over 24 months, the investigators will examine all patients diagnosed with proctosigmoiditis at the Department of Liver, Digestive, and Gastrointestinal Diseases at Aarhus University Hospital (AUH), Viborg/Silkeborg Regional Hospital, Horsens Regional Hospital, Gødstrup Regional Hospital and Randers Regional Hospital. This includes patients with inflammation extending from the anal opening to 35 cm proximally, as well as those with treatment-refractory proctosigmoiditis.

All patient data will be prospectively collected through Region Midt EPJ, Denmark's electronic medical record system, and registered in a REDCap database.

The tested patients will undergo standard follow-up at their respective departments. Supple-mentary, patients who test positive for Chlamydia or Gonorrhoea will be offered treatment at the Venereology Outpatient Clinic, Aarhus University Hospital. If they are only on 5-ASA treatment and it is found reasonable to pause their treatment, their IBD treatment will be paused during treatment for STI.

The studied patients will form a prospective cohort, and their disease progression, including the extent of haemorrhagic proctitis and current medication, will be recorded.

Endpoints

Primary endpoint:

- Prevalence of Chlamydia and Gonorrhoea in our cohort of individuals with suspected haemorrhagic proctitis.

Secondary endpoints:

* Prevalence of Chlamydia and Gonorrhoea across gender
* Prevalence of Chlamydia and Gonorrhoea across age groups
* Prevalence of Chlamydia and Gonorrhoea depending on time for diagnosis
* Frequency of clinical remission of proctitis after treatment with STI-related antibiotics
* Differences in the frequency of clinical remission between those with a negative or positive STI test at inclusion

DETAILED DESCRIPTION:
Protocol The prevalence of Chlamydia trachomatis and Neisseria gonorrhoeae in patients suspected of hemorrhagic proctosigmoiditis (SOS Proctitis)

A quality improvement project in the Central Denmark Region

Background Chlamydia trachomatis and Neisseria gonorrhoeae can cause infectious proctitis, which macroscopically cannot be distinguished from haemorrhagic proctosigmoiditis (HP) caused by inflammatory bowel disease. In Denmark, general practitioners are advised to consider whether patients presenting with proctitis symptoms might have a sexually transmitted infection (STI). However, there is no requirement for STI testing before referring the patient to a specialised department.

At specialised departments, it is not standard of care to systematically inquire about sexual risk behaviour or to test for Chlamydia and Gonorrhoea. As a result, there is no data on how many patients diagnosed with HP due to chronic inflammatory bowel disease are also positive for an STI, either as the sole cause or as a contributing factor to their inflammation. Chlamydia and Gonorrhoea are the most common causes of symptomatic, sexually transmitted proctitis and are increasingly prevalent in Denmark.

Aims To investigate the proportion of patients with newly diagnosed proctosigmoiditis or treatment-refractory disease who have an underlying STI, to determine whether the prevalence of STIs varies across sex or age groups, while also investigating whether STIs are prevalent in both newly diagnosed patients and patients with refractory disease, and to monitor the effect of antibiotic treatment on proctitis progression. The implications of these findings could help determine whether screening for these pathogens should be implemented as part of the standard diagnostic process for haemorrhagic proctosigmoiditis.

Materials and methods Since diagnosing haemorrhagic proctosigmoiditis requires an endoscopy (sigmoidoscopy or colonoscopy), all newly diagnosed patients will undergo such an examination. Moreover, an endoscopy is often performed in individuals with refractory proctosigmoiditis. If inflammation is observed up to 35 cm from the anal verge, an additional swab will be taken during the procedure to test for Chlamydia and Gonorrhoea using standard PCR techniques. If the swab is not taken during the endoscopy, it will be collected during a follow-up outpatient visit. The tests will be analysed immediately at the Department of Microbiology, Aarhus University Hospital.

Over 24 months, all patients diagnosed with proctosigmoiditis at the Department of Liver, Digestive, and Gastrointestinal Diseases at Aarhus University Hospital (AUH), Viborg/Silkeborg Regional Hospital, Horsens Regional Hospital, Gødstrup Regional Hospital and Randers Regional Hospital will be offered a rectal swab. This includes patients with inflammation extending from the anal opening to 35 cm proximally, as well as those with treatment-refractory proctosigmoiditis.

All patient data will be prospectively collected through Region Midt EPJ, Denmark's electronic medical record system, and registered in a REDCap database.

The tested patients will undergo standard follow-up at their respective departments. Supplementary, patients who test positive for Chlamydia or Gonorrhoea will be offered treatment at the Venereology Outpatient Clinic, Aarhus University Hospital. If they are only on 5-ASA treatment and it is found reasonable to pause their treatment, their IBD treatment will be paused during treatment for STI.

The studied patients will form a prospective cohort, and their disease progression, including the extent of haemorrhagic proctitis and current medication, will be recorded.

Endpoints

Primary endpoint:

- Prevalence of Chlamydia and Gonorrhoea in our cohort of individuals with suspected haemorrhagic proctitis.

Secondary endpoints:

* Prevalence of Chlamydia and Gonorrhoea across gender
* Prevalence of Chlamydia and Gonorrhoea across age groups
* Prevalence of Chlamydia and Gonorrhoea depending on time for diagnosis
* Frequency of clinical remission of proctitis after treatment with STI-related antibiotics
* Differences in the frequency of clinical remission between those with a negative or positive STI test at inclusion

Statistical analysis The statistical analyses will mainly be descriptive. For the primary and secondary outcomes, numbers with frequencies will be reported. Furthermore, appropriate statistical analyses will be applied to compare differences between those with a positive STI test and those with a negative test.

The data collection period runs from October 1, 2024, until September 30, 2026, and we expect to include at least 100 patients in the cohort, but aim towards at least 200 patients. After 100 patients have been tested, it will be assessed whether it is feasible to continue to screen patients. If no positive patients have been found, the study will terminate prematurely. By September 2025, it will be evaluated whether to publish the results before 200 unique participants have been included; this will be considered if more than 5% of all patients examined are positive or if an isolated group has a more than 15% positive rate.

The results will be submitted for publication regardless of the outcome.

Ethical considerations To assess whether screening for STI in patients suspected of HP should be mandatory, screening for STI in patients suspected of HP has become a recommended clinical procedure in Region Midt in the current study period. All patients will give oral consent to perform the swab during the endoscopy or in the outpatient ward. Local authorities have approved the collection of data for a quality improvement project.

Perspectives If Chlamydia and Gonorrhea are found frequently, these results could indicate the necessity for integrating screening practices for all newly diagnosed HP patients and those with treatment-refractory disease.

If patients improve after pathogen-directed treatment and avoid treatment-refractory disease, there could be cost reduction if fewer biological therapies and patient visits are required.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected of haemorrhagic proctosigmoiditis with either newly diagnosed or recurrent disease who undergo lower endoscopy

Exclusion Criteria:

* Patients who does not accept the swap to be taken

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suspected of haemorrhagic proctosigmoiditis with either newly diagnosed or recurrent disease who undergo lower endoscopy
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Chlamydia in individuals with suspected haemorrhagic proctitis | 2 years
  Number of Chlamydia positive individuals on rectal swap
Prevalence of Gonorrhoea in individuals with suspected haemorrhagic proctitis | 2 years
  Number of Gonorrhoea positive individuals on rectal swap

SECONDARY OUTCOMES:
Prevalence of Chlamydia across gender | 2 years
Prevalence Gonorrhoea across gender | 2 years
Prevalence of Chlamydia across age groups | 2 years
Prevalence of Gonorrhoea across age groups | 2 years
Prevalence of Chlamydia depending on time for diagnosis | 2 years
  Defined whether the individual has debut of HP at the time of positive test, or refractory disease
Prevalence of Gonorrhoea depending on time for diagnosis | 2 years
  Defined whether the individual has debut of HP at the time of positive test, or refractory disease
Frequency of clinical remission of proctitis after treatment with STI-related antibiotics | 2 years
  8 and 12 weeks after antibiotic treatment
Differences in the frequency of clinical remission between those with a negative or positive STI test at inclusion | 2 years
  8 and 12 weeks after antibiotic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christan L Hvass, Professor, Study Chair — Aarhus University Hospital; Line Kibsgaard, MD, Ph.D., Study Chair — Aarhus University Hospital; Anders K Dige, Consultant, Ph.D., Principal Investigator — Aarhus University Hospital
Locations (5):
- Denmark (5):
  - Aarhus University Hospital, Aarhus N
  - Gødstrup Regional Hospital, Herning
  - Randers Regional Hospital, Randers
  - Silkeborg Regional Hospital, Silkeborg
  - Viborg Regional Hospital, Viborg

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be shared beginning 9 months and ending 36 months foliowing article publication.
Access Criteria: Data will be shared to researchers who provide a methodologically sound proposal and have been approved by the principal investigator.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Clinical trials protocol (2025-04-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT07061899/Prot_SAP_000.pdf
  • Study Protocol: Inital internal protocol (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT07061899/Prot_001.pdf